CLINICAL TRIAL: NCT04875728
Title: Evaluating the Impact of Perioperative Antibiotic Prophylaxis on the Microbiome in Patients With Cutaneous Malignancy
Brief Title: The Impact of an Antibiotic (Cefazolin) Before Surgery on the Microbiome in Patients With Stage I-II Melanoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0265; NCI-2020-07071 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0265 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-05; First posted 2021-05-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Clinical Stage I Cutaneous Melanoma AJCC v8; Clinical Stage IA Cutaneous Melanoma AJCC v8; Clinical Stage IB Cutaneous Melanoma AJCC v8; Clinical Stage II Cutaneous Melanoma AJCC v8; Clinical Stage IIA Cutaneous Melanoma AJCC v8; Clinical Stage IIB Cutaneous Melanoma AJCC v8; Clinical Stage IIC Cutaneous Melanoma AJCC v8; Pathologic Stage I Cutaneous Melanoma AJCC v8; Pathologic Stage IA Cutaneous Melanoma AJCC v8; Pathologic Stage IB Cutaneous Melanoma AJCC v8; Pathologic Stage II Cutaneous Melanoma AJCC v8; Pathologic Stage IIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIC Cutaneous Melanoma AJCC v8
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (cefazolin, surgical resection) (Active Comparator): Patients receive cefazolin IV and then undergo standard of care surgical resection within 1 hour.
  Interventions: Drug: Cefazolin; Procedure: Resection
- Arm B (surgical resection) (Experimental): Patients undergo standard of care surgical resection.
  Interventions: Procedure: Resection

INTERVENTIONS:
Drug: Cefazolin — Given IV
  Arms: Arm A (cefazolin, surgical resection)
Procedure: Resection — Undergo standard of care surgical resection
  Other Names: Surgical Resection

SUMMARY:
This phase I trial investigates the impact of cefazolin before surgery on the microbiome in patients with stage I-II melanoma. Antibiotics, such as cefazolin, given at the time of surgery may cause a significant change in the microbes (like bacteria and viruses) found in the stomach and intestines. This trial may help researchers learn if any changes in microbes affect the body's ability to respond to surgery and cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate whether the use of pre-operative prophylactic antibiotics administered during surgical resection substantially alters the patient's gut microbiome.

SECONDARY OBJECTIVES:

I. To characterize the dynamics of the immune response to surgical intervention in the absence and presence of pre-operative prophylactic antibiotics, focusing on the immune profile of the peripheral blood leukocytes as well as the balance of circulating pro- and anti-inflammatory cytokines and metabolomic profiles.

II. To assess surgical site infection (SSI) in the absence and presence of pre-operative prophylactic antibiotics at time of surgical resection.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive cefazolin intravenously (IV) and then undergo standard of care surgical resection within 1 hour.

ARM B: Patients undergo standard of care surgical resection.

After completion of study treatment, patients are followed up at 3 days, 2 weeks, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with early stage melanoma (stage I-II)
* Patients must be undergoing wide local excision +/- sentinel lymph node biopsy
* Patients must be capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* Use of antibiotics within the three months prior to surgery
* Allergy, sensitivity or anaphylaxis to beta-lactam or cephalosporin antibiotics
* Presence of an infection at the time of surgery
* Increased risk of infection due to a co-existing medical condition as determined by the surgical team or principal investigator (PI)
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration
* American Society of Anesthesiologists (ASA) grade > IV
* Refusal to participate in the study
* Patients who are pregnant will not be included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in microbiome alpha diversity | Baseline up to 2 weeks post-surgery
  The diversity, structure, and composition of the fecal microbiome will be determined by 16S(v4) rRNA gene sequencing. 16S profiles will be used to compute alpha diversity, beta diversity, and the relative abundance of fecal bacteria. The composition of fecal bacteria in adult humans is mainly dominated by members of the Firmicutes and Proteobacteria phyla while members of Proteobacteria, Actinobacteria, Fusobacteria, and Verrucomicrobia are observed in lower abundance. To calculate richness (alpha-diversity), we will count each operational taxonomic unit (OTU) or amplicon sequence variant (ASV) identified. Richness count is expected to range between 10-500 per sample.

SECONDARY OUTCOMES:
Change in relative abundance of microbes | Baseline, at 2 weeks post-surgery, and 3 months post-surgery
Change in microbiome diversity | Baseline up to 3 months post-surgery
  The diversity, structure, and composition of the fecal microbiome will be determined by 16S(v4) rRNA gene sequencing. 16S profiles will be used to compute alpha diversity, beta diversity, and the relative abundance of fecal bacteria. The composition of fecal bacteria in adult humans is mainly dominated by members of the Firmicutes and Proteobacteria phyla while members of Proteobacteria, Actinobacteria, Fusobacteria, and Verrucomicrobia are observed in lower abundance. To calculate richness (alpha-diversity), we will count each operational taxonomic unit (OTU) or amplicon sequence variant (ASV) identified. Richness count is expected to range between 10-500 per sample.
Wound (surgical site) infection rate | Up to 3 months post-surgery
Profiling of systemic immune function by analysis of composition of circulating immune cell populations and cytokines | Up to 3 months post-surgery
  By analysis of composition of circulating immune cell populations and cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Z Keung, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT04875728/ICF_000.pdf